CLINICAL TRIAL: NCT01919944
Title: A Randomized, Double-Blind, Placebo-Controlled, Four-Way Crossover Study on Itch Control by VLY-686 Administration in Healthy Volunteers After Intradermal Injections of Substance P
Brief Title: Study of Itch Control by VLY-686 in Healthy Volunteers After Intradermal Injections of Substance P
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VP-VLY-686-1101
Record Dates: First submitted 2013-08-02; First posted 2013-08-09 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Pruritus
Keywords: itch
MeSH Terms: conditions — Pruritus | interventions — LY686017

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- VLY-686 20 mg (Experimental): Single dose, 20 mg VLY-686, administered as two 10 mg VLY-686 oral capsules
  Interventions: Drug: VLY-686
- VLY-686 50 mg (Experimental): Single dose, 50 mg VLY-686, administered as one 50 mg VLY-686 oral capsule and one placebo capsule mimicking the VLY-686 50 mg capsule
  Interventions: Drug: VLY-686; Drug: Placebo
- VLY-686 100 mg (Experimental): Single dose, 100 mg VLY-686, administered as two 50 mg VLY-686 oral capsules
  Interventions: Drug: VLY-686
- Placebo (Placebo Comparator): Single dose, placebo, administered as either two 10 mg oral capsules or two 50 mg oral capsules
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VLY-686 — capsules containing either 10 mg or 50 mg VLY-686
  Arms: VLY-686 100 mg; VLY-686 20 mg; VLY-686 50 mg
Drug: Placebo — Sugar capsule to mimic either VLY-686 10 mg capsule or 50 mg capsule
  Arms: Placebo; VLY-686 50 mg

SUMMARY:
The purpose of this study is to test whether VLY-686 can prevent or reduce the itch and dermatological reaction observed after healthy volunteers are injected with Substance P in comparison with placebo.

DETAILED DESCRIPTION:
This is a double-blind, randomized, 4-way crossover, pharmacokinetic and pharmacodynamic (PK/PD) study to compare the cutaneous vasoreactive intensity to intradermal injections of Substance P in healthy volunteers receiving oral doses of 20 mg, 50 mg or 100 mg VLY-686 or a matching placebo. Twelve healthy male subjects satisfying the selection criteria for the study will be enrolled. Each subject will participate in a screening period (up to 21 days prior to dosing), four one-day treatment periods each separated by a 7 (±2 days) day washout period, and an end-of-study evaluation prior to discharge from the study. This protocol also includes an option of subjects administered daily doses of study medication between Periods 3 and 4. The treatment periods will be in a randomized sequence consisting of 1) 20 mg VLY-686, 2) 50 mg VLY-686, 100 mg VLY-686 and 4) placebo. In each of the study periods, Substance P will be injected 5 times: pre-dose (the night before), 2, 4, 8 and 12 hours (± 10 minutes) after study medication administration. A dose of 100 μL of a 2.5 nmol/mL sterile solution of Substance P will be injected each time. Overall, subjects will be administered 1.25 nmol of Substance P in around 24 hours (5 doses). Substance P injections will be given in the volar of the forearm, alternating right and left and avoiding injections in an area adjacent to the area previously injected. The subject's forearm will be covered during and after each injection to avoid potential biases in the scoring of the Verbal Rating Scale (VRS) and Visual Analog Scale (VAS). Additionally, blood samples for VLY-686 pharmacokinetic (PK) analysis will be collected each period at pre-dose, 1, 3, 6, 10, and 24 hours after study medication administration.

ELIGIBILITY:
Inclusion Criteria:

* Males 18 - 45 years of age, inclusive;
* Non-smokers, per medical history, or ex-smokers for a period of ≥1 year;
* Subjects with Body Mass Index (BMI) of ≥18.5 and ≤30 kg/m2 (BMI = weight (kg)/ [height (m)]2);
* Vital signs (in sitting position after 3 minutes of rest) which are within the ranges shown below (inclusive):
* Body temperature between 35.4-37.8 °C;
* Systolic blood pressure between 91-130 mmHg;
* Diastolic blood pressure between 51-90 mmHg;
* Pulse rate between 50-100 bpm;
* Respiratory rate between 10-20 breaths per minute;
* Ability and acceptance to provide written informed consent;
* Willing and able to comply with study requirements and restrictions;
* Subjects must be in good health as determined by past medical history, physical examination, electrocardiogram, clinical laboratory tests and urinalysis.

Exclusion Criteria:

* Past or present history of atopy (atopic dermatitis problems, urticaria, asthma or allergic rhinitis) with no ascertained intolerance to histamine;
* Past or present skin disease;
* Lesions or any skin changes in the forearms in the month prior to the Screening Visit;
* History of neurological diseases;
* Past or present pain-related diseases such as cluster headaches, migraine, or back pain;
* Treatment with all topical cream and ointments including cosmetics applied on the forearm in the 10 days prior to the screening visit;
* Participation in the evaluation of any investigational product for 3 months before this study, calculated from the first day of the month following the last visit of the previous study;
* Exposure (within 2 weeks of the Baseline Visit) to any prescription medication or over-the-counter medication including dietary supplements and/or herbal remedies, except those listed on Section 8.2;
* Exposure (within 4 weeks of the Screening Visit) to any antihistamines, anxiolytics, antidepressants, pain killers including triptanes, neuroleptics, or sleep medications;
* Treatment with any medication known to cause major organ system toxicity (e.g., chloramphenicol or tamoxifen) during the 60 days preceding the Screening Visit;
* Administration of medications containing corticosteroids or adrenocorticotropic hormone in the three months prior to the Screening Visit;
* Electrocardiogram reading considered outside the normal limits by the investigator (e.g. abnormally prolonged QTc corrected by Fridericia's method > 450 msec in males, on ECG tracing). The following conduction abnormalities may confound QTc analysis and should be avoided if possible: PR > 220 msec, 2nd or 3rd degree AV block, intraventricular conduction delay with QRS > 120 msec, left branch bundle block, right branch bundle block or Wolff-Parkinson-White syndrome;
* Blood donation in the last 3 months or donation of at least 1500 mL blood (including this study) within the last year;
* History of liver disease and/or positive for one or more of the following serological results:
* A positive hepatitis C antibody test (anti-HCV);
* A positive hepatitis B surface antigen (HBsAg);
* A positive HIV test result ;
* Not willing to sign the informed consent or not able to understand completely the study objectives or risks;
* Clinically relevant abnormalities in clinical lab or physical assessments performed at the screening visit;
* Lack of sensitivity to Substance P and histamine or sensitivity to saline at the Screening Visit;
* Any other sound medical reason as determined by the clinical Investigator.
* Drug, alcohol, caffeine, tobacco: history of drug, alcohol (>2 drinks/day for males, defined according to USDA Dietary Guidelines 2010), caffeine (>5 cups coffee/tea/day), smokers;
* Diet: abnormal diets (<1600 or >3500 calories/day) or substantial changes in eating habits in the 4 weeks before this study; vegetarians.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2013-08; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Itch severity score on the Verbal Rating Scale | 20 minutes after Substance P injection
Itch severity score on the Visual Analog Scale | 20 minutes after Substance P injection

SECONDARY OUTCOMES:
Dose response of VLY-686 and reduction of itch severity | 20 minutes after substance P injection
Number of adverse events in subjects taking VLY-686 | 24 hours after Substance P injection
Size of injection site erythema | 1-20 minutes after Substance P injection
Number of adverse events in subjects taking placebo | 20 minutes after Substance P inection
Size of injection site and urticaria | 20 minutes after Substance P injection

CONTACTS AND LOCATIONS:
Overall Officials: Milko Radicioni, MD, Principal Investigator — Cross Research SA
Locations (1):
- Vanda Investigational Site, Arzo, Switzerland